CLINICAL TRIAL: NCT03013205
Title: Efficacy of Corticosteroid Injection Into Coracohumeral Ligament in Patients With Adhesive Capsulitis of the Shoulder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201609026RINB
Record Dates: First submitted 2016-12-26; First posted 2017-01-06 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Direct Coracohumeral Ligament Steroid Injection
Keywords: adhesive capsulitis
MeSH Terms: conditions — Bursitis | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- PT+IA+CHL (Experimental): 1. Intraarticular triamcinolone injection
  2. Intraarticular Xylocaine injection
  3. Coracohumeral ligament triamcinolone injection
  4. Physiotherapy
  Interventions: Procedure: Intraarticular triamcinolone injection; Procedure: Intraarticular Xylocaine injection; Procedure: Coracohumeral ligament triamcinolone injection; Procedure: Physiotherapy
- PT+IA (Active Comparator): 1. Intraarticular triamcinolone injection
  2. Intraarticular Xylocaine injection
  3. Physiotherapy
  Interventions: Procedure: Intraarticular triamcinolone injection; Procedure: Intraarticular Xylocaine injection; Procedure: Physiotherapy

INTERVENTIONS:
Procedure: Intraarticular triamcinolone injection — triamcinolone 10mg/mL
Procedure: Intraarticular Xylocaine injection — Xylocaine 1% 4ml
Procedure: Coracohumeral ligament triamcinolone injection — triamcinolone 10mg/mL
  Arms: PT+IA+CHL
Procedure: Physiotherapy

SUMMARY:
Steroid injections are widely utilized to reduce inflammation and fibrosis in patients with the frozen shoulder. In this study, investigators will compare intra-articular steroid injections with direct coracohumeral ligament steroid injection to conventional intra-articular steroid injection. Investigators will measure the primary outcome as shoulder function improvement and secondary outcomes as ROM, pain scale and stiffness of coracohumeral ligament under elastogram.

DETAILED DESCRIPTION:
Adhesive capsulitis of the shoulder, also known as the frozen shoulder, often leads to severe pain and shoulder range of motion limitation. Steroid injections are widely utilized to reduce inflammation and fibrosis. The thickening of the coracohumeral ligament was thought to play an important role in the pathogenesis of frozen shoulder, resulting in limited external rotation of the shoulder. While the elastogram of coracohumeral ligament will significantly increase stiffness under the shear-wave ultrasound (shear-wave elastography).

Therefore, in this study, investigators will compare intra-articular steroid injections with direct coracohumeral ligament steroid injection to conventional intra-articular steroid injection. Investigators will measure the primary outcome as shoulder function improvement and secondary outcomes as ROM, pain scale and stiffness of coracohumeral ligament under elastogram.

(the patient will not have additional risk of injection under ultrasound guidance)

ELIGIBILITY:
A.Inclusion criteria：

1. Age 20-80 years old
2. Unilateral shoulder pain more than 3 months
3. At least one shoulder ROM limitation in three dimensions which decreased over 50% (Abduction, Flexion, External rotation)
4. Visual analog scale more than 30 (total 100)
5. No fracture or subluxation or arthritis in shoulder Xray.

B.Exclusion criteria：

1. History of shoulder or chest surgery
2. History of shoulder trauma in 2 recent years
3. Ever receiving shoulder joint injection in recent 3 months
4. With cervical radiculopathy or any central CNS disorders
5. With osteoarthritis or rheumatic arthritis of shoulder
6. Diagnosed as rotator cuff tear, tendon calcification or bursitis
7. Systemic diseases including diabetes or thyroid disorder
8. Allergy history of steroid

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-02; Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Shoulder function (The Disabilities of the Arm, Shoulder and Hand Score, QuickDash) improvement | 2 years
  shoulder function improvement (The Disabilities of the Arm, Shoulder and Hand Score, QuickDash), score 0-100

SECONDARY OUTCOMES:
Change of Visual analogue scale | 2 years
  Visual analogue scale: scale 0-10
Shoulder range of motion improvement | 2 years
  Range of motion improvement: flexion, abduction, external rotation (degree)
Stiffness of coracohumeral ligament under elastogram (KPa) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Chueh-Hung Wu, MD, Principal Investigator — NTUH PMR
Locations (1):
- National Taiwan University Hospital, Test1, Test2, Taiwan